CLINICAL TRIAL: NCT05967832
Title: Contribution of 7 Tesla MRI of the Hypothalamus in the Diagnosis of Type 1 Narcolepsy: Pilot Study
Brief Title: Contribution of 7 Tesla MRI of the Hypothalamus in the Diagnosis of Type 1 Narcolepsy
Acronym: NARCO7T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM22_0378; ID-RCB (Other: 2022-A02674-39)
Record Dates: First submitted 2023-04-23; First posted 2023-08-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Narcolepsy Type 1
Keywords: narcolepsy; 7T MRI; hypothalamus
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with type 1 narcolepsy (Experimental): Patients with type 1 narcolepsy
  Interventions: Other: 7T MRI
- Healthy volunteers (Active Comparator)
  Interventions: Other: 7T MRI

INTERVENTIONS:
Other: 7T MRI — Patients and healthy volunteers will have a 7T MRI

SUMMARY:
This study is part of the research on type 1 narcolepsy, a neurological pathology affecting mostly young subjects. The only biomarker currently available is the hypocretin assay, which shows a level below 110 pg/mL. However, the interpretation of this biomarker has limitations: the test is not widely available and it is rarely performed by practitioners. Even when performed, the interpretation of the level may not be consistent with the phenotype compatible with type 1 narcolepsy.

This study therefore aims to develop new tools to reduce the diagnostic delay. This would be the first study with 7T MRI that could achieve a level of spatial resolution sufficient to highlight volume changes in small brain structures such as the lateral hypothalamus whose narcolepsy-induced changes are not detected by lower resolution MRI.

ELIGIBILITY:
Inclusion Criteria for patients :

1. Diagnosis of narcolepsy type 1 according to the diagnostic criteria of the International Classification of sleep disorders version 3 (ICSD-3, American Academy of Sleep Medicine, 2014) including a mean sleep latency of less than 8 minutes on the iterative sleep latency test associated with at least two direct REM sleep onset and the presence of cataplexy, and a cerebrospinal fluid hypocretin assay of less than 110 pg/ml performed by the reference radioimmunology (RIA) technique.
2. Patient at least 18 years old
3. Patient followed at the Narcolepsy and Rare Hypersomnias Competence Center, Timone Hospital, Marseille
4. Patient having signed an informed consent
5. Patient who is a beneficiary of or affiliated to a social security system

Exclusion Criteria for patient:

1. Diagnosis of type 1 narcolepsy according to ICSD-3 criteria but without hypocretin assay
2. Narcolepsy secondary to another neurological pathology or presence of a comorbid neurological pathology (multiple sclerosis, Steinert's myotonic dystrophy, head trauma, epilepsy)
3. Protected patient: pregnant or breastfeeding woman, adult under guardianship or curatorship
4. Contraindication to the realization of a 7T MRI: patient wearing a pacemaker, neurosurgical clips, artificial heart valve, surgical material or metal fragments in the body, dental or hearing prostheses, insulin pump, patient wearing an IUD, claustrophobic patient
5. Patient unable to maintain decubitus position for the duration of the MRI (= 50 minutes)

Inclusion criteria for healthy volunteers:

1. Subject 18 years of age or older
2. Subject free of general illness, psychiatric disorders, and infectious, inflammatory, tumor, vascular, degenerative, or traumatic pathology of the central nervous system as determined during the medical interview.
3. Subject who has signed an informed consent ;
4. Subjects who are beneficiaries of or affiliated with a social security plan

Exclusion criteria for healthy volunteers:

1. Protected subject: pregnant or breastfeeding woman, adult under guardianship or curatorship
2. Subjects presenting a contraindication to the realization of a 7T MRI: patient with a pacemaker, neurosurgical clips, artificial heart valve, surgical material or metal fragments in the body, dental or auditory prostheses, insulin pump, patient with an IUD, claustrophobic patient
3. Subject unable to maintain a decubitus position for the duration of the MRI (= 50 minutes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Hypothalamic morphological difference | Month 0
  Significant structural size difference between right and left lateral hypothalamus

SECONDARY OUTCOMES:
Microstructural abnormalities other than volume differences | Month 0
  Significant difference in Diffusion and T2* values in the lateral hypothalamus
Structural changes in hypothalamic nuclei other than the lateral hypothalamus | Month 0
  Significant difference in volumes and T1 values in other regions of the posterior hypothalamus

CONTACTS AND LOCATIONS:
Overall Officials: François Crémieux, Study Director — AP-HM
Locations (1):
- Service Epileptologie et Rythmologie Cérébrale, Centre du Sommeil, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided